CLINICAL TRIAL: NCT07163156
Title: The Relationship of Prolactin and Inflammatory Markers With Parkinson's Disease Severity: Clinical and Biochemical Evaluation
Brief Title: Prolactin, Inflammation, and Parkinson's Severity
Acronym: PRIPS
Status: Enrolling by invitation | Type: Observational
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Hüseyin Avni Eroğlu, Assoc. Prof., Çanakkale Onsekiz Mart University
Other Study IDs: COMU-FNN-1; NOT YET (Other Grant/Funding Number: Canakkale Onsekiz Mart University)
Record Dates: First submitted 2025-08-23; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Idiopathic Parkinson Disease; Prolactin; Prolactin Levels; Inflammation
MeSH Terms: conditions — Parkinson Disease; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Parkinson's Disease Patients

SUMMARY:
This cross-sectional observational study aims to evaluate the relationship between serum prolactin levels, peripheral inflammatory markers (NLR, PLR, SII, CRP), and disease severity in patients with Parkinson's disease (PD). A total of at least 300 patients diagnosed with idiopathic PD will be included. Disease severity will be assessed using the Unified Parkinson's Disease Rating Scale (UPDRS) and the Modified Hoehn-Yahr staging system. Serum and salivary prolactin levels will be measured using ELISA, while inflammatory markers will be calculated from routine blood tests. The study seeks to clarify whether prolactin and systemic inflammation indicators may serve as non-invasive biomarkers for disease progression and prognosis in PD, with particular emphasis on postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of idiopathic Parkinson's disease confirmed by a neurologist
* Both male and postmenopausal female patients
* Patients able to provide informed consent
* Clinically stable enough to undergo blood and saliva sampling, as well as neurological assessment

Exclusion Criteria:

* Premenopausal female patients
* Patients with secondary or atypical parkinsonism (e.g., drug-induced, vascular, atypical parkinsonian syndromes)
* Known endocrine disorders affecting prolactin levels (e.g., prolactinoma, pituitary adenoma, hypothyroidism)
* Use of medications known to alter prolactin secretion (e.g., antipsychotics, dopamine antagonists, estrogen therapy)
* History of other neurodegenerative diseases (e.g., Alzheimer's, Huntington's)
* Presence of active infection, chronic inflammatory disease, or malignancy
* Severe renal, hepatic, or cardiac failure
* Inability to provide informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of at least 300 adult patients (≥18 years) diagnosed with idiopathic Parkinson's disease who are followed at the Neurology Department of Çanakkale Onsekiz Mart University. Both male and postmenopausal female patients will be included. Participants must be clinically stable and able to undergo neurological evaluation, serum and salivary prolactin testing, and routine laboratory investigations. Patients with atypical or secondary parkinsonism, endocrine disorders affecting prolactin levels, active infection, chronic inflammatory disease, or malignancy will be excluded.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Systemic inflammatory markers | 1 year later
  NLR, PLR, SII, CRP
Prolactin Level | 1 year later
  Serum prolactine levels

CONTACTS AND LOCATIONS:
Locations (1):
- Çanakkale Onsekiz Mart University, Çanakkale, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided